CLINICAL TRIAL: NCT03306446
Title: Changing the coUrse of cRohn's Disease With an Early Use of Adalimumab
Acronym: CURE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2013-1
Record Dates: First submitted 2015-06-21; First posted 2017-10-11 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: CD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab in monotherapy (Experimental): Start Adalimumab in monotherapy at 160 mg at inclusion, 80 mg on 2nd week and 40 mg/week each other week over 12 months.
  Interventions: Drug: Start adalimumab in monotherapy

INTERVENTIONS:
Drug: Start adalimumab in monotherapy — Discontinuation of Adalimumab in patients who achieved deep remission
  Other Names: begin humira in monotherapie in Early crohn disease patient

SUMMARY:
This is a prospective, longitudinal, multicenter study conducted in a cohort of patients with early CD. This study will not change the patient/physician relationship.

DETAILED DESCRIPTION:
The main objective will be to evaluate the sustained deep remission rate one year after discontinuation of a 12 month course of adalimumab in adult patients with early CD who have achieved deep remission at 12 months AND who were already in clinical remission (CDAI < 150) and biomarker remission (CRP < 5 mg/L and fecal calprotectin < 250) at 6 months. The study will also address several questions:

* What is the rate of deep remission after a 12-month course of adalimumab in early CD patients?
* What is the rate of deep remission 12 months after adalimumab discontinuation in patients with deep remission after a 12-month course of adalimumab (thus defining sustained deep remission) AND who were already in clinical remission (CDAI < 150) and biomarker remission (CRP < 5 mg/L and fecal calprotectin < 250) at 6 months?
* What are the consequences of a treatment with adalimumab on the natural course of CD and long-term clinical outcomes (bowel damage, CD related surgeries and hospitalization, and patient-reported outcomes)? Therefore the study will give information on the effect of a 12-month course of adalimumab in early CD patients, impact of "drug holiday" after deep remission has been achieved, and long term effect of adalimumab on early CD course (relapses, CD-related surgery and hospitalizations, bowel damage, and patient-reported outcomes). The study will also assess predictors of loss of deep remission at 2-year evaluation in patients who achieved 1-year deep remission. Efficacy and tolerability of adalimumab will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years old to 75 years old 2. Patient with early luminal Crohn's disease (less than 24 months since diagnosis), 3. Patient who is
* intolerant to immunosuppressants or steroids, or
* primarily not responders to immunosuppressants for at least 3 months [azathioprine: at least 2.5 mg/kg/d; 6-mercaptopurine: at least 1.5 mg/kg/d; methotrexate: 25 mg/week (subcutaneous or intramuscular route)], and/or
* not responder to steroids [prednisolone equivalent at least 40 mg/d], and/or
* steroid-dependent [unable to reduce corticosteroids below the equivalent of prednisolone 10 mg/d or budesonide < 6 mg/d within 3 months of starting corticosteroids without recurrent active disease, or who have a relapse within 3 months of stopping corticosteroids], 4. Patient with CDAI > 150, 5. Patient with at least one ulcer in at least one affected segment (Magnetic Resonance Imaging (MRI) of gastrointestinal tract or colonoscopy or by video capsule conducted after failure of conventional therapy and within 12 weeks before inclusion in the study), 6. Patient naïve for anti-TNF, 7. Patient whose physician decides to start adalimumab as monotherapy independently from the study protocol, 8. Patient followed in a centre belonging to the GETAID network. 9. Written consent.

Exclusion Criteria:

* Patient with active complex perianal fistula according to the definition of the American Gastroenterological Association (AGA) [high anal fistula, abscess, proctitis, multiple external openings],
* Patient with stoma,
* previous surgery in IBD
* Pregnant or breastfeeding women, absence of contraception
* Patient with any contra-indication to adalimumab.
* Patient with any contra-indication to MRI
* Minors and people unable to give their consent (because of their physical or mental state).
* Subject who has not given his/her consent to participate.
* Subject participating in another study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Sustained deep remission rate | 12 months
  Number of patients with sustained deep remission at one year

SECONDARY OUTCOMES:
2-year deep remission rate | 2 years
  Number of patients with 2-year deep remission rate among patients who did not achieve 1-year remission

OTHER OUTCOMES:
Impact of an early treatment with adalimumab on long-term clinical outcomes | 5 years
  Frequency and severity of adverse events in patients followed for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Bouhnik, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Laurent Peyrin-Biroulet, MD, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (23):
- Chu Liege, Liège, Belgium
- France (22):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - CHU de Caen- Hopital de la Cote de Nacre, Caen
  - CHU de CLERMONT FERRAND- Hopital Estain, Clermont-Ferrand
  - APHP- Hopital BEAUJON, Clichy
  - CHU de Colmar- Hopital Trousseau Medecine A, Colmar
  - Chu Lille, Lille
  - CHU de Montpellier- Hopital saint Eloi, Montpellier
  - CHU NANTES - Hôpital Hôtel Dieu, Nantes
  - CHU de NICE- Hopital Archet 2, Nice
  - CHU de Nimes- Hopital Carémeau, Nîmes
  - APHP- Hopital COCHIN, Paris
  - APHP- Hopital BICHAT, Paris
  - IMM, Paris
  - CHU Bordeaux- Hopital Haut Levèque, Pessac
  - CHU LYON- Hopital Lyon Sud, Pierre-Bénite
  - CHU RENNES - Hopital Pontchaillou, Rennes
  - CHU de Saint Etienne- Hopital Nord, Saint-Priest-en-Jarez
  - CHU de TOULOUSE, Toulouse
  - CHU de Tours - Hopital Trousseau, Tours
  - CH Valenciennes, Valenciennes
  - CHU NANCY - Hopital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided